CLINICAL TRIAL: NCT01465763
Title: A Multicentre, Randomized, Double-blind, Placebo-controlled, Parallel-group Study Of Oral Cp-690,550 As An Induction Therapy In Subjects With Moderate To Severe Ulcerative Colitis
Brief Title: A Study Evaluating The Efficacy And Safety Of CP-690,550 In Patients With Moderate To Severe Ulcerative Colitis
Acronym: OCTAVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3921094; 2011-004578-27 (EudraCT Number); OCTAVEINDUCTION1 (Other: Alias Study Number)
Record Dates: First submitted 2011-10-21; First posted 2011-11-07 (Estimated); Results first posted 2016-06-07 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-05

CONDITIONS: Ulcerative Colitis
Keywords: tofacitinib; CP-690; 550; Moderate to severe ulcerative colitis; phase 3 clinical trial; Mayo score
MeSH Terms: conditions — Colitis, Ulcerative | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tofacitinib 10 mg BID (Experimental)
  Interventions: Drug: tofacitinib
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: tofacitinib — 10 mg oral BID
  Other Names: CP-690,550
  Arms: tofacitinib 10 mg BID
Drug: Placebo — Plabebo oral BID
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the efficacy and safety of tofacitinib (CP-690,550) in patients with moderate to severe ulcerative colitis who have failed or be intolerant to one of following treatments for ulcerative colitis: oral steroids, azathiopurine/6-mercaptopurine, or anti-TNF-alpha therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age.
* Males and females with a documented diagnosis of UC at least 4 months prior to entry into the study.
* Subjects with moderately to severely active UC based on Mayo score criteria.
* Subjects must have failed or be intolerant of at least one of the following treatments for UC:

  * Corticosteroids (oral or intravenous).
  * Azathioprine or 6 mercaptopurine (6 MP).
  * Anti TNF-alpha therapy.

Exclusion Criteria:

* Presence of indeterminate colitis, microscopic colitis, ischemic colitis, infectious colitis, or clinical findings suggestive of Crohn's disease.
* Subjects with disease limited to distal 15 cm.
* Subjects without previous treatment for UC (ie, treatment naïve).
* Subjects displaying clinical signs of fulminant colitis or toxic megacolon.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 2012-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (178):
- United States (71):
  - Internal Medicine Center, LLC, Mobile, Alabama
  - Springhill Memorial Hospital, Mobile, Alabama
  - Investigational Drug Service Pharmacy, La Jolla, California
  - UCSD Medical Center, La Jolla, California
  - UCSD Medical Centre, La Jolla, California
  - Cedars Sinai Medical Center - Thalians Bldg, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Cedars Sinai Surgery Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - CRC Office - Cedars-Sinai Medical Center - Inflammatory Bowel Disease Center, Los Angeles, California
  - Desert Advanced Imaging, Palm Springs, California
  - Erik Palmer, DO, Palm Springs, California
  - Homan A Zadeh, MD, MPH, Palm Springs, California
  - Hope Square Surgical Center, Rancho Mirage, California
  - Sharp Rees-Stealy Medical Group, Inc., San Diego, California
  - Sharp Rees-Stealy Medical Group, San Diego, California
  - Sharp Rees-Stealy Medical Group,Inc, San Diego, California
  - Endoscopy Center of Connecticut, LLC, Guilford, Connecticut
  - Endoscopy Center of Connecticut, LLC, Hamden, Connecticut
  - Gastroenterology Center of Connecticut, PC, Hamden, Connecticut
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - Florida Surgery Center, Altamonte Springs, Florida
  - Center for Advanced Gastroenterology, Maitland, Florida
  - MNH Surgical Center, Maitland, Florida
  - Sand Lake Imaging, Maitland, Florida
  - North Florida Gastroenterology Research, LLC, Orange Park, Florida
  - Orange Park Surgery Center, Orange Park, Florida
  - Citrus Ambulatory Surgery Center, Orlando, Florida
  - Internal Medicine Specialists, Orlando, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Florida Medical Clinic, P.A., Zephyrhills, Florida
  - Georgia Endoscopy Center (Colonoscopy only), Alpharetta, Georgia
  - GI Consultants (Colonoscopy only), Atlanta, Georgia
  - Emory Healthcare Heart Center (EKG), Johns Creek, Georgia
  - Gastroenterology Associates of Central Georgia, Macon, Georgia
  - Icahn School of Medicine at Mount Sinai, Marietta, Georgia
  - Atlanta Gastroenterology Specialists, PC, Suwanee, Georgia
  - Johns Creek Diagnostic Center (X-Ray only), Suwanee, Georgia
  - Southwest Gastroenterology, Oak Lawn, Illinois
  - Saint Joseph Mercy Hospital - Inpatient Pharmacy (Pharmacy Only), Ann Arbor, Michigan
  - East Ann Arbor Health and Geriatrics Center - University of Michigan Health Systems, Ann Arbor, Michigan
  - University of Michigan Health Systems, Ann Arbor, Michigan
  - Michigan Clinical Research Unit - Univeristy of Michigan Health System, Ann Arbor, Michigan
  - Medical Science Research Building 1 - University of Michigan Health Systems, Ann Arbor, Michigan
  - Michigan Heart SJMH (Blood draws and ECGs only), Ypsilanti, Michigan
  - Huron Gastroenterology Associates / Center for Digestive Care, Ypsilanti, Michigan
  - Saint Joseph Mercy Hospital Outpatient Laboratory (Blood draws only), Ypsilanti, Michigan
  - Center for Advanced Medicine, St Louis, Missouri
  - Washington University School of Medicine - Division of Gastroenterology, St Louis, Missouri
  - NYU Langone Long Island Clinical Research Associates, Great Neck, New York
  - NYU Langone Nassau Gastroenterology Associates, Great Neck, New York
  - The Private Practice of Simon Lichtiger, MD, New York, New York
  - Mount Sinai Doctos Faculty Practice, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - CUMC Research Pharmacy, New York, New York
  - Kornbluth, Legnani, George MD, PC, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Great Lakes Gastroenterology, Mentor, Ohio
  - Mentor Medical Campus, Mentor, Ohio
  - The Endoscopy Center of Lake County, Mentor, Ohio
  - Houston Hospital for Specialized Surgery, Houston, Texas
  - Baylor College of Medicine (Baylor Medical Center), Houston, Texas
  - Baylor College of Medicine - Baylor Medical Center (Drug Storage), Houston, Texas
  - Gastroenterology Consultants, P.A., Houston, Texas
  - Alpine Medical Group, Salt Lake City, Utah
  - Wasatch Clinical Research, Salt Lake City, Utah
  - Wasatch Endoscopy Center, Salt Lake City, Utah
  - RGL Medical Services (x-ray only), West Jordan, Utah
  - Wisconsin Center for Advanced Research - GI Associates, LLC, Milwaukee, Wisconsin
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Eastern Health Box Hill Hospital, Box Hill, Victoria
- AKH Wien, Universitaetsklinik fuer Innere Medizin III,, Vienna, Austria
- UZ Leuven (University Hospital Leuven), Campus Gasthuisberg, Leuven, Belgium
- Canada (5):
  - Hertiage Medical Research Clinic- University Of Calgary, Calgary, Alberta
  - McMaster University Medical Center, Hamilton, Ontario
  - Hamilton Health Sciences Corporation - McMaster University Medical Centre, Hamilton, Ontario
  - London Health Sciences Centre - University Hospital, London, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
- Unidad de Gastroenterologia y Endoscopia Digestiva S.A. - UGASEND S.A., Barranquilla, Atlántico, Colombia
- General Hospital Zadar, Zadar, Croatia
- Czechia (3):
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - Institut klinicke a experimentalni mediciny, Prague
  - Klinicke Centrum ISCARE I.V.F., Prague
- Denmark (2):
  - Aalborg Hospital, Aalborg
  - Aarhus University Hospital, Aarhus C
- Estonia (3):
  - ECG Unit of West Tallinn Central Hospital, Tallinn
  - West Tallinn Central Hospital Internal Diseases Clinic, Tallinn
  - X-Ray Department of West Tallinn Central Hospital, Tallinn
- France (3):
  - CHU de Nantes - Hotel Dieu, Nantes
  - Hopital Saint-Louis, Paris
  - Hopital Rangueil, Toulouse
- Germany (4):
  - Universitaetsmedizin Berlin, Charite Campus Virchow-Klinikum,, Berlin
  - Universitaetsklinikum Halle (Saale), Halle
  - Medizinische Hochschule Hannover, Hanover
  - Klinikum Luneburg/Abteilung Gastroenterologie, Lüneburg
- Hungary (4):
  - Szent Margit Korhaz III Belgyogyaszati Gasztroenterologiai Osztaly, Budapest
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
  - Szegedi Tudomanyegyetem Altalanos Orvostudomanyi Kar I. sz. Belgyogyaszati Klinika, Szeged
  - Javorszky Odon Korhaz/Gasztroenterologiai Osztaly, Vác
- Israel (2):
  - Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
  - Rabin Medical Center, Beilinson campus, Petah Tikva
- Italy (6):
  - AOU Mater Domini - U.O. Fisiopatologia Digestiva, Catanzaro, CZ
  - Istituto Clinico Humanitas IRCSS, Rozzano, Milano
  - IBD Center - IRCCS Humanitas, Milan, Milan
  - A.O.R. Villa Sofia- Cervello, Palermo, PA
  - Comitato Etico Palermo 2, Palermo, PA
  - SOC Gastroenterologia Centro di Riferimento Oncologico, Aviano
- Japan (23):
  - Aichi Medical University Hospital, Nagakute, Aichi-ken
  - National Hospital Organization Hirosaki National Hospital, Hirosaki, Aomori
  - Chiba University Hospital, Chiba, Chiba
  - Toho University Sakura Medical Center, Sakura, Chiba
  - Kurume University Hospital, Kurume, Fukuoka
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Hokkaido P.W.F.A.C Sapporo-Kosei general Hospital, Sapporo, Hokkaido
  - The Hospital of Hyogo College of Medicine, Nishinomiya, Hyōgo
  - National Hospital Organization Mito Medical Center, Higashi-ibaraki-gun, Ibaraki
  - Kuniyoshi Hospital, Kochi, Kochi
  - National Hospital Organization Sendai Medical Center, Sendai, Miyagi
  - Osaka City University Hospital, Osaka, Osaka
  - Osaka Medical College Hospital, Takatsuki-shi, Osaka
  - Shiga University of Medical Science Hospital, Ōtsu, Shiga
  - Tokai University Hachioji Hospital, Hachiōji, Tokyo
  - Jikei University Hospital, Minato-ku, Tokyo
  - Kitasato University Kitasato Institute Hospital, Minato-ku, Tokyo
  - NTT Medical Center Tokyo, Shinagawa-ku, Tokyo
  - Showa University Hospital, Shinagawa-ku, Tokyo
  - Keio University Hospital, Tokyo, Tokyo
  - Fukuoka University Chikushi Hospital, Fukuoka
  - Sameshima Hospital, Kagoshima
  - Tokyo Medical And Dental University Hospital, Faculty of Medicine, Tokyo
- Latvia (3):
  - Digestive Diseases Center GASTRO, Riga
  - ECG room, Clinic "Linezers", Riga
  - X-Ray Department, Clinic "Linezers", Riga
- Leiden University Medical Center, Leiden, South Holland, Netherlands
- New Zealand (3):
  - Shakespeare Specialist Group, Milford, Auckland
  - Southern District Health Board, Dunedin
  - Bop Clinical School Clinical Trials Unit, Tauranga
- Poland (4):
  - Gabinet Lekarski - Janusz Rudzinski, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Klinika Chorob Wewnetrznych i Gastroenterologii z Pododdzialem Leczenia, Warsaw, Masovian Voivodeship
  - Oddzial Kliniczny Gastroenterologii Ogolnej i Onkologicznej SP ZOZ Uniwersytecki, Lodz
  - Lexmedica, Wroclaw
- Cabinet Particular Policlinic Algomed SRL, Timișoara, Jud Timis, Romania
- Russia (11):
  - Municipal budget institution of healthcare "Central City Hospital of Pyatigorsk", Pyatigorsk, Stavropol Kray
  - State budgetInstitution ofHealthcare Nizhniy NovgorodRegionalClinicalHospital namedafterN.A.Semashko, Nizhny Novgorod
  - Federal State Institution "Sibirian regional Medical Centre of Federal Medicobiologic Agency", Novosibirsk
  - Municipal budget institution of healthcare of Novosibirsk "City Clinical Hospital, Novosibirsk
  - State Budget Educational Institution of Higher Professional Education, Novosibirsk
  - Federal State Budgetary Military Educational Institution of High Professional Education, Saint Petersburg
  - GBOU VPO "Northwest State Medical University n.a. I.I. Mechnikov", Saint Petersburg
  - GUZ City Hospital #26, Saint Petersburg
  - Non-State Healthcare Institution "Road Clinical Hispital at the station Samara" of Open Joint-Stock, Samara
  - Limited Liability Company Medical Company "Hepatolog", Samara
  - Samara Diagnostic center, X-ray Department, Samara
- Serbia (4):
  - General Hospital "Djordje Joanovic" Department for Gastroenterology and Hepatology, Zrenjanin, Serbia, Europe
  - Clinical Hospital Centre Zvezdara, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Centre of Kragujevac, Kragujevac
- Medak s.r.o., Bratislava, Slovakia, Slovakia
- South Africa (2):
  - Chris Hani Baragwanath Academic Hospital, Johannesburg, Gauteng
  - Endocare Research Centre, Cape Town, Western Cape
- Spain (4):
  - Hospital Clinico San Carlos, Madrid, Madrid
  - Hospital Clínic i provincial de Barcelona, Barcelona
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario de Fuenlabrada, Madrid
- Ukraine (9):
  - InternalMedicineCenterofCrimean RepublicInstitution"ClinicalTerritorialMedicalCommunity"University, Simferopol, Ar Krym
  - State Institution "National L.T. Malaya Therapy Institute of National Academy, Kharkiv, Ukraine
  - Kyiv Municipal Clinical Hospital #18, Proctology Department, Kyiv
  - LTD "St. Paraskeva Medical Center", Lviv
  - Municipal City Clinical Hospital of the Emergency Medical Care, 1-st Therapy Department of hospital,, Lviv
  - SI "Railway Hospital of the SI "Odesa Railway"", Polyclinic Department,, Odesa
  - SI "District Clin. Hosp.of Uzhgorod station (STSA "Lviv Railway", Therapy Dep., SBHEI, Uzhhorod
  - Vinnytsia National Medical University, Vinnytsia
  - Vinnytsia Regional Clinical Hospital for Invalids of the Great Patriotic War, Therapy Department #2, Vinnytsia
- United Kingdom (2):
  - Cambridge University Hospitals Nhs Foundation Trust, Cambridge
  - University College London Hospital, London

REFERENCES:
- [Derived] Rubin DT, Torres J, Regueiro M, Reinisch W, Prideaux L, Kotze PG, Tan FH, Gardiner S, Mundayat R, Cadatal MJ, Ng SC. Association Between Smoking Status and the Efficacy and Safety of Tofacitinib in Patients with Ulcerative Colitis. Crohns Colitis 360. 2024 Jan 20;6(1):otae004. doi: 10.1093/crocol/otae004. eCollection 2024 Jan. PMID 38425446
- [Derived] Rubin DT, Salese L, Cohen M, Kotze PG, Woolcott JC, Su C, Mundayat R, Paulissen J, Torres J, Long MD. Presence of risk factors associated with colectomy among patients with ulcerative colitis: a post hoc analysis of data from the tofacitinib OCTAVE ulcerative colitis clinical program. Therap Adv Gastroenterol. 2023 Aug 7;16:17562848231189122. doi: 10.1177/17562848231189122. eCollection 2023. PMID 37560161
- [Derived] Schreiber S, Rubin DT, Ng SC, Peyrin-Biroulet L, Danese S, Modesto I, Guo X, Su C, Kwok KK, Jo H, Chen Y, Yndestad A, Reinisch W, Dubinsky MC. Major Adverse Cardiovascular Events by Baseline Cardiovascular Risk in Patients with Ulcerative Colitis Treated with Tofacitinib: Data from the OCTAVE Clinical Programme. J Crohns Colitis. 2023 Nov 24;17(11):1761-1770. doi: 10.1093/ecco-jcc/jjad104. PMID 37402275
- [Derived] Kristensen LE, Danese S, Yndestad A, Wang C, Nagy E, Modesto I, Rivas J, Benda B. Identification of two tofacitinib subpopulations with different relative risk versus TNF inhibitors: an analysis of the open label, randomised controlled study ORAL Surveillance. Ann Rheum Dis. 2023 Jul;82(7):901-910. doi: 10.1136/ard-2022-223715. Epub 2023 Mar 17. PMID 36931693
- [Derived] Lichtenstein GR, Cohen BL, Salese L, Modesto I, Wang W, Chan G, Ahmed HM, Su C, Peyrin-Biroulet L. Impact of Concomitant Corticosteroids on Tofacitinib Induction Efficacy and Infection Rates in Ulcerative Colitis. Dig Dis Sci. 2023 Jun;68(6):2624-2634. doi: 10.1007/s10620-022-07794-0. Epub 2023 Feb 4. PMID 36739367
- [Derived] Dubinsky MC, Armuzzi A, Gecse KB, Ullman T, Bushmakin AG, DiBonaventura M, Cappelleri JC, Connelly SB, Woolcott JC, Salese L. Improvements in Disease Activity Partially Mediate the Effect of Tofacitinib Treatment on Generic and Disease-Specific Health-Related Quality of Life in Patients with Ulcerative Colitis: Data from the OCTAVE Program. Dig Dis. 2023;41(4):604-614. doi: 10.1159/000528788. Epub 2023 Jan 5. PMID 36603566
- [Derived] Winthrop KL, Yndestad A, Henrohn D, Danese S, Marsal S, Galindo M, Woolcott JC, Jo H, Kwok K, Shapiro AB, Jones TV, Diehl A, Su C, Panes J, Cohen SB. Influenza Adverse Events in Patients with Rheumatoid Arthritis, Ulcerative Colitis, or Psoriatic Arthritis in the Tofacitinib Clinical Development Programs. Rheumatol Ther. 2023 Apr;10(2):357-373. doi: 10.1007/s40744-022-00507-z. Epub 2022 Dec 17. PMID 36526796
- [Derived] Sandborn WJ, Sands BE, Vermeire S, Leung Y, Guo X, Modesto I, Su C, Wang W, Panes J. Modified Mayo score versus Mayo score for evaluation of treatment efficacy in patients with ulcerative colitis: data from the tofacitinib OCTAVE program. Therap Adv Gastroenterol. 2022 Dec 5;15:17562848221136331. doi: 10.1177/17562848221136331. eCollection 2022. PMID 36506749
- [Derived] Lichtenstein GR, Bressler B, Francisconi C, Vermeire S, Lawendy N, Salese L, Sawyerr G, Shi H, Su C, Judd DT, Jones T, Loftus EV. Assessment of Safety and Efficacy of Tofacitinib, Stratified by Age, in Patients from the Ulcerative Colitis Clinical Program. Inflamm Bowel Dis. 2023 Jan 5;29(1):27-41. doi: 10.1093/ibd/izac084. PMID 36342120
- [Derived] Hudesman DP, Torres J, Salese L, Woolcott JC, Mundayat R, Su C, Mosli MH, Allegretti JR. Long-Term Improvement in the Patient-Reported Outcomes of Rectal Bleeding, Stool Frequency, and Health-Related Quality of Life with Tofacitinib in the Ulcerative Colitis OCTAVE Clinical Program. Patient. 2023 Mar;16(2):95-103. doi: 10.1007/s40271-022-00603-w. Epub 2022 Nov 7. PMID 36336750
- [Derived] Targownik L, Dubinsky MC, Steinwurz F, Bushmakin AG, Cappelleri JC, Tai E, Gardiner S, Hur P, Panes J. Disease Activity and Health-related Quality of Life Relationships with Work Productivity in Patients with Ulcerative Colitis in OCTAVE Induction 1 and 2 and OCTAVE Sustain. J Crohns Colitis. 2023 Apr 19;17(4):513-523. doi: 10.1093/ecco-jcc/jjac161. PMID 36271912
- [Derived] Sandborn WJ, D'Haens GR, Sands BE, Panaccione R, Ng SC, Lawendy N, Kulisek N, Modesto I, Guo X, Mundayat R, Su C, Vranic I, Panes J. Tofacitinib for the Treatment of Ulcerative Colitis: An Integrated Summary of up to 7.8 Years of Safety Data from the Global Clinical Programme. J Crohns Colitis. 2023 Apr 3;17(3):338-351. doi: 10.1093/ecco-jcc/jjac141. PMID 36124702
- [Derived] Loftus EV, Baumgart DC, Gecse K, Kinnucan JA, Connelly SB, Salese L, Su C, Kwok KK, Woolcott JC, Armuzzi A. Clostridium difficile Infection in Patients with Ulcerative Colitis Treated with Tofacitinib in the Ulcerative Colitis Program. Inflamm Bowel Dis. 2023 May 2;29(5):744-751. doi: 10.1093/ibd/izac139. PMID 35792493
- [Derived] Winthrop KL, Vermeire S, Long MD, Panes J, Ng SC, Kulisek N, Mundayat R, Lawendy N, Vranic I, Modesto I, Su C, Melmed GY. Long-term Risk of Herpes Zoster Infection in Patients With Ulcerative Colitis Receiving Tofacitinib. Inflamm Bowel Dis. 2023 Jan 5;29(1):85-96. doi: 10.1093/ibd/izac063. PMID 35648151
- [Derived] Mukherjee A, Tsuchiwata S, Nicholas T, Cook JA, Modesto I, Su C, D'Haens GR, Sandborn WJ. Exposure-Response Characterization of Tofacitinib Efficacy in Moderate to Severe Ulcerative Colitis: Results From Phase II and Phase III Induction and Maintenance Studies. Clin Pharmacol Ther. 2022 Jul;112(1):90-100. doi: 10.1002/cpt.2601. Epub 2022 Apr 27. PMID 35380740
- [Derived] Dubinsky MC, Magro F, Steinwurz F, Hudesman DP, Kinnucan JA, Ungaro RC, Neurath MF, Kulisek N, Paulissen J, Su C, Ponce de Leon D, Regueiro M. Association of C-reactive Protein and Partial Mayo Score With Response to Tofacitinib Induction Therapy: Results From the Ulcerative Colitis Clinical Program. Inflamm Bowel Dis. 2023 Jan 5;29(1):51-61. doi: 10.1093/ibd/izac061. PMID 35380664
- [Derived] Feagan BG, Khanna R, Sandborn WJ, Vermeire S, Reinisch W, Su C, Salese L, Fan H, Paulissen J, Woodworth DA, Niezychowski W, Sands BE. Agreement between local and central reading of endoscopic disease activity in ulcerative colitis: results from the tofacitinib OCTAVE trials. Aliment Pharmacol Ther. 2021 Dec;54(11-12):1442-1453. doi: 10.1111/apt.16626. Epub 2021 Oct 6. PMID 34614208
- [Derived] Farraye FA, Qazi T, Kotze PG, Moore GT, Mundayat R, Lawendy N, Sharma PP, Judd DT. The impact of body mass index on efficacy and safety in the tofacitinib OCTAVE ulcerative colitis clinical programme. Aliment Pharmacol Ther. 2021 Aug;54(4):429-440. doi: 10.1111/apt.16439. Epub 2021 Jun 24. PMID 34165201
- [Derived] Rubin DT, Reinisch W, Greuter T, Kotze PG, Pinheiro M, Mundayat R, Maller E, Fellmann M, Lawendy N, Modesto I, Vavricka SR, Lichtenstein GR. Extraintestinal manifestations at baseline, and the effect of tofacitinib, in patients with moderate to severe ulcerative colitis. Therap Adv Gastroenterol. 2021 May 16;14:17562848211005708. doi: 10.1177/17562848211005708. eCollection 2021. PMID 34035832
- [Derived] Sandborn WJ, Peyrin-Biroulet L, Sharara AI, Su C, Modesto I, Mundayat R, Gunay LM, Salese L, Sands BE. Efficacy and Safety of Tofacitinib in Ulcerative Colitis Based on Prior Tumor Necrosis Factor Inhibitor Failure Status. Clin Gastroenterol Hepatol. 2022 Mar;20(3):591-601.e8. doi: 10.1016/j.cgh.2021.02.043. Epub 2021 Mar 6. PMID 33684552
- [Derived] Vong C, Martin SW, Deng C, Xie R, Ito K, Su C, Sandborn WJ, Mukherjee A. Population Pharmacokinetics of Tofacitinib in Patients With Moderate to Severe Ulcerative Colitis. Clin Pharmacol Drug Dev. 2021 Mar;10(3):229-240. doi: 10.1002/cpdd.899. Epub 2021 Jan 29. PMID 33513294
- [Derived] Curtis JR, Regueiro M, Yun H, Su C, DiBonaventura M, Lawendy N, Nduaka CI, Koram N, Cappelleri JC, Chan G, Modesto I, Lichtenstein GR. Tofacitinib Treatment Safety in Moderate to Severe Ulcerative Colitis: Comparison of Observational Population Cohort Data From the IBM MarketScan(R) Administrative Claims Database With Tofacitinib Trial Data. Inflamm Bowel Dis. 2021 Aug 19;27(9):1394-1408. doi: 10.1093/ibd/izaa289. PMID 33324993
- [Derived] Sandborn WJ, Peyrin-Biroulet L, Quirk D, Wang W, Nduaka CI, Mukherjee A, Su C, Sands BE. Efficacy and Safety of Extended Induction With Tofacitinib for the Treatment of Ulcerative Colitis. Clin Gastroenterol Hepatol. 2022 Aug;20(8):1821-1830.e3. doi: 10.1016/j.cgh.2020.10.038. Epub 2020 Oct 27. PMID 33127596
- [Derived] Sands BE, Colombel JF, Ha C, Farnier M, Armuzzi A, Quirk D, Friedman GS, Kwok K, Salese L, Su C, Taub PR. Lipid Profiles in Patients With Ulcerative Colitis Receiving Tofacitinib-Implications for Cardiovascular Risk and Patient Management. Inflamm Bowel Dis. 2021 May 17;27(6):797-808. doi: 10.1093/ibd/izaa227. PMID 32870265
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Dubinsky MC, DiBonaventura M, Fan H, Bushmakin AG, Cappelleri JC, Maller E, Thorpe AJ, Salese L, Panes J. Tofacitinib in Patients with Ulcerative Colitis: Inflammatory Bowel Disease Questionnaire Items in Phase 3 Randomized Controlled Induction Studies. Inflamm Bowel Dis. 2021 Jun 15;27(7):983-993. doi: 10.1093/ibd/izaa193. PMID 32794567
- [Derived] Lichtenstein GR, Rogler G, Ciorba MA, Su C, Chan G, Pedersen RD, Lawendy N, Quirk D, Nduaka CI, Thorpe AJ, Panes J. Tofacitinib, an Oral Janus Kinase Inhibitor: Analysis of Malignancy (Excluding Nonmelanoma Skin Cancer) Events Across the Ulcerative Colitis Clinical Program. Inflamm Bowel Dis. 2021 May 17;27(6):816-825. doi: 10.1093/ibd/izaa199. PMID 32766762
- [Derived] Sandborn WJ, Panes J, Sands BE, Reinisch W, Su C, Lawendy N, Koram N, Fan H, Jones TV, Modesto I, Quirk D, Danese S. Venous thromboembolic events in the tofacitinib ulcerative colitis clinical development programme. Aliment Pharmacol Ther. 2019 Nov;50(10):1068-1076. doi: 10.1111/apt.15514. Epub 2019 Oct 9. PMID 31599001
- [Derived] Sands BE, Taub PR, Armuzzi A, Friedman GS, Moscariello M, Lawendy N, Pedersen RD, Chan G, Nduaka CI, Quirk D, Salese L, Su C, Feagan BG. Tofacitinib Treatment Is Associated With Modest and Reversible Increases in Serum Lipids in Patients With Ulcerative Colitis. Clin Gastroenterol Hepatol. 2020 Jan;18(1):123-132.e3. doi: 10.1016/j.cgh.2019.04.059. Epub 2019 May 8. PMID 31077827
- [Derived] Sandborn WJ, Panes J, D'Haens GR, Sands BE, Su C, Moscariello M, Jones T, Pedersen R, Friedman GS, Lawendy N, Chan G. Safety of Tofacitinib for Treatment of Ulcerative Colitis, Based on 4.4 Years of Data From Global Clinical Trials. Clin Gastroenterol Hepatol. 2019 Jul;17(8):1541-1550. doi: 10.1016/j.cgh.2018.11.035. Epub 2018 Nov 23. PMID 30476584
- [Derived] Hanauer S, Panaccione R, Danese S, Cheifetz A, Reinisch W, Higgins PDR, Woodworth DA, Zhang H, Friedman GS, Lawendy N, Quirk D, Nduaka CI, Su C. Tofacitinib Induction Therapy Reduces Symptoms Within 3 Days for Patients With Ulcerative Colitis. Clin Gastroenterol Hepatol. 2019 Jan;17(1):139-147. doi: 10.1016/j.cgh.2018.07.009. Epub 2018 Sep 10. PMID 30012431
- [Derived] Winthrop KL, Melmed GY, Vermeire S, Long MD, Chan G, Pedersen RD, Lawendy N, Thorpe AJ, Nduaka CI, Su C. Herpes Zoster Infection in Patients With Ulcerative Colitis Receiving Tofacitinib. Inflamm Bowel Dis. 2018 Sep 15;24(10):2258-2265. doi: 10.1093/ibd/izy131. PMID 29850873
- [Derived] Motoya S, Watanabe M, Kim HJ, Kim YH, Han DS, Yuasa H, Tabira J, Isogawa N, Arai S, Kawaguchi I, Hibi T. Tofacitinib induction and maintenance therapy in East Asian patients with active ulcerative colitis: subgroup analyses from three phase 3 multinational studies. Intest Res. 2018 Apr;16(2):233-245. doi: 10.5217/ir.2018.16.2.233. Epub 2018 Apr 30. PMID 29743836
- [Derived] Panes J, Vermeire S, Lindsay JO, Sands BE, Su C, Friedman G, Zhang H, Yarlas A, Bayliss M, Maher S, Cappelleri JC, Bushmakin AG, Rubin DT. Tofacitinib in Patients with Ulcerative Colitis: Health-Related Quality of Life in Phase 3 Randomised Controlled Induction and Maintenance Studies. J Crohns Colitis. 2018 Jan 24;12(2):145-156. doi: 10.1093/ecco-jcc/jjx133. PMID 29028981
- [Derived] Sandborn WJ, Su C, Sands BE, D'Haens GR, Vermeire S, Schreiber S, Danese S, Feagan BG, Reinisch W, Niezychowski W, Friedman G, Lawendy N, Yu D, Woodworth D, Mukherjee A, Zhang H, Healey P, Panes J; OCTAVE Induction 1, OCTAVE Induction 2, and OCTAVE Sustain Investigators. Tofacitinib as Induction and Maintenance Therapy for Ulcerative Colitis. N Engl J Med. 2017 May 4;376(18):1723-1736. doi: 10.1056/NEJMoa1606910. PMID 28467869
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921094&StudyName=A%20Study%20Evaluating%20The%20Efficacy%20And%20Safety%20Of%20CP-690%2C550%20In%20Patients%20With%20Moderate%20To%20Severe%20Ulcerative%20Colitis

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to tofacitinib 10 milligram (mg) or placebo twice a day (BID)(4:1 ratio) after protocol amendment 3, which removed tofacitinib 15 mg BID. Due to low participant numbers, tofacitinib 15 mg BID was excluded from efficacy analyses, but was included in participant flow, baseline characteristics and adverse events analyses.
Groups:
- Tofacitinib 10 mg BID: Participants received tofacitinib 10 mg, tablets, orally, BID for 9 weeks of double blind treatment period.
- Tofacitinib 15 mg BID: Participants received tofacitinib 15 mg, tablets, orally, BID for 9 weeks of double blind treatment period.
- Placebo BID: Participants received tofacitinib-matched placebo tablets, orally, BID for 9 weeks of double blind treatment period.
Period: Overall Study
Arm/Group | Tofacitinib 10 mg BID | Tofacitinib 15 mg BID | Placebo BID
Started | 476 | 16 | 122
Completed | 445 | 15 | 118
Not Completed | 31 | 1 | 4
Not completed — Withdrawal by Subject | 4 | 0 | 1
Not completed — Insufficient Clinical Response | 11 | 0 | 1
Not completed — Adverse Event | 9 | 0 | 1
Not completed — Other | 2 | 0 | 0
Not completed — Protocol Violation | 4 | 1 | 1
Not completed — Death | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set consists of all randomized participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tofacitinib 10 mg BID | Tofacitinib 15 mg BID | Placebo BID | Total
Number analyzed (Participants) | 476 | 16 | 122 | 614
Age, Customized [Number; unit: participants]
  18 to 44 Years | 295 | 11 | 72 | 378
  45 to 64 Years | 145 | 4 | 39 | 188
  Greater Than or Equal to (>=) 65 Years | 36 | 1 | 11 | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 199 | 7 | 45 | 251
  Male | 277 | 9 | 77 | 363

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Remission at Week 8
Description: Remission in participants was defined by a total Mayo score of 2 points or lower, with no individual subscore exceeding 1 point and a rectal bleeding subscore of 0. Mayo score is an instrument designed to measure disease activity of ulcerative colitis (UC). It consisted of 4 subscores: stool frequency, rectal bleeding, findings of centrally read flexible proctosigmoidoscopy and physician global assessment (PGA), each graded from 0 to 3 with higher scores indicating more severe disease. These scores were summed up to give a total score range of 0 to 12; where higher scores indicating more severe disease.
Time Frame: Week 8
Population: Full analysis set (FAS) included all participants randomly assigned to either tofacitinib 10 mg BID or placebo BID.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 476 | 122
percentage of participants | 18.5 | 8.2
Statistical Analysis 1: Comparison: Tofacitinib 10 mg BID vs Placebo BID; P-value based on Cochran-Mantel-Haenszel (CMH) chi-square test stratified by prior treatment with anti-tumor necrosis factor (TNF), steroid use at baseline and geographic region. Difference and its 95% CI based on normal approximation for the difference in binomial proportions. Missing data were imputed using Non-responder imputation (NRI); Test type: Superiority or Other; p = 0.0070, CMH Chi-square test; Percent Difference = 10.3, 95% CI 2-sided [4.3 to 16.3]

2. Secondary Outcome: Percentage of Participants Achieving Mucosal Healing at Week 8
Description: Mucosal healing in participants was defined by Mayo endoscopic subscore of 0 or 1. The Mayo endoscopic subscore consisted of the findings of centrally read flexible proctosigmoidoscopy, graded from 0 to 3 with higher scores indicating more severe disease.
Time Frame: Week 8
Population: FAS included all participants randomly assigned to either tofacitinib 10 mg BID or placebo BID.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 476 | 122
percentage of participants | 31.3 | 15.6
Statistical Analysis 1: Comparison: Tofacitinib 10 mg BID vs Placebo BID; P-value based on CMH chi-square test stratified by prior treatment with anti-TNF, steroid use at baseline and geographic region. Difference and its 95% CI based on normal approximation for the difference in binomial proportions. Missing data were imputed using NRI; Test type: Superiority or Other; p = 0.0005, CMH Chi-square test; Percent Difference = 15.7, 95% CI 2-sided [8.1 to 23.4]

3. Secondary Outcome: Percentage of Participants Achieving Clinical Response at Week 8
Description: Clinical response in participants was defined by a decrease from baseline in Mayo score of at least 3 points and at least 30 percent, with an accompanying decrease in the rectal bleeding subscore of at least 1 point or an absolute rectal bleeding subscore of 0 or 1. Mayo score is an instrument designed to measure disease activity of UC. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of centrally read flexible proctosigmoidoscopy and PGA, each graded from 0 to 3 with higher scores indicating more severe disease. These scores were summed up to give a total score range of 0 to 12; where higher scores indicating more severe disease.
Time Frame: Week 8
Population: FAS included all participants randomly assigned to either tofacitinib 10 mg BID or placebo BID.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 476 | 122
percentage of participants | 59.9 | 32.8
Statistical Analysis 1: Comparison: Tofacitinib 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, CMH Chi-square test; Percent Difference = 27.1, 95% CI 2-sided [17.7 to 36.5]

4. Secondary Outcome: Percentage of Participants With Endoscopic Remission at Week 8
Description: Endoscopic remission in participants was defined by Mayo endoscopic subscore of 0. The Mayo endoscopic subscore consisted of the findings of centrally read flexible proctosigmoidoscopy, graded from 0 to 3 with higher scores indicating more severe disease.
Time Frame: Week 8
Population: FAS included all participants randomly assigned to either tofacitinib 10 mg BID or placebo BID.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 476 | 122
percentage of participants | 6.7 | 1.6
Statistical Analysis 1: Comparison: Tofacitinib 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0345, CMH Chi-square test; Percent Difference = 5.1, 95% CI 2-sided [1.9 to 8.3]

5. Secondary Outcome: Percentage of Participants With Clinical Remission at Week 8
Description: Clinical remission in participants was defined by a total Mayo score of 2 points or lower, with no individual subscore exceeding 1 point. Mayo score is an instrument designed to measure disease activity of UC. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of centrally read flexible proctosigmoidoscopy and PGA, each graded from 0 to 3 with higher scores indicating more severe disease. These scores were summed up to give a total score range of 0 to 12; where higher scores indicating more severe disease.
Time Frame: Week 8
Population: FAS included all participants randomly assigned to either tofacitinib 10 mg BID or placebo BID.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 476 | 122
percentage of participants | 18.5 | 8.2
Statistical Analysis 1: Comparison: Tofacitinib 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0070, CMH Chi-square test; Percent Difference = 10.3, 95% CI 2-sided [4.3 to 16.3]

6. Secondary Outcome: Percentage of Participants With Symptomatic Remission at Week 8
Description: Symptomatic remission in participants was defined by a total Mayo score of 2 points or lower, with no individual subscore exceeding 1 point, and 0 subscore for both rectal bleeding and stool frequency. Mayo score is an instrument designed to measure disease activity of UC. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of centrally read flexible proctosigmoidoscopy and PGA, each graded from 0 to 3 with higher scores indicating more severe disease. These scores were summed up to give a total score range of 0 to 12; where higher scores indicating more severe disease.
Time Frame: Week 8
Population: FAS included all participants randomly assigned to either tofacitinib 10 mg BID or placebo BID.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 476 | 122
percentage of participants | 11.8 | 5.7
Statistical Analysis 1: Comparison: Tofacitinib 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0601, CMH Chi-square test; Percent Difference = 6.0, 95% CI 2-sided [1.0 to 11.1]

7. Secondary Outcome: Percentage of Participants With Deep Remission at Week 8
Description: Deep remission in participants was defined by a total Mayo score of 2 points or lower, with no individual subscore exceeding 1 point and 0 subscore for both rectal bleeding and endoscopic subscores. Mayo score is an instrument designed to measure disease activity of UC. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of centrally read flexible proctosigmoidoscopy and PGA, each graded from 0 to 3 with higher scores indicating more severe disease. These scores were summed up to give a total score range of 0 to 12; where higher scores indicating more severe disease.
Time Frame: Week 8
Population: FAS included all participants randomly assigned to either tofacitinib 10 mg BID or placebo BID.
Measure: Number; unit: percentage of participants
Arm/Group | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 476 | 122
percentage of participants | 6.5 | 0
Statistical Analysis 1: Comparison: Tofacitinib 10 mg BID vs Placebo BID; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0043, CMH Chi-square test; Percent Difference = 6.5, 95% CI 2-sided [4.3 to 8.7]

8. Secondary Outcome: Partial Mayo Scores
Description: A Partial Mayo Score (mayo score without endoscopy) graded from 0 (normal or inactive disease) to 9 (severe disease) and calculated as the sum of 3 subscores (stool frequency, rectal bleeding and PGA) with each grading from 0 to 3 with higher scores indicating more severe disease.
Time Frame: Baseline, Weeks 2, 4, 8
Population: FAS included all participants randomly assigned to either tofacitinib 10 mg BID or placebo BID. Here, 'n' signifies those participants who were evaluable at specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 476 | 122
units on a scale
  Baseline: (n= 475, 121) | 6.3 (1.2) | 6.5 (1.2)
  At Week 2: (n= 465, 122) | 4.2 (2.2) | 5.2 (2.1)
  At Week 4: (n= 461, 118) | 3.5 (2.3) | 4.8 (2.4)
  At week 8: (n= 449, 119) | 3.2 (2.4) | 4.8 (2.5)

9. Secondary Outcome: Change From Baseline in Partial Mayo Scores at Weeks 2, 4 and 8
Description: Change in partial mayo scores at weeks 2, 4, 8 relative to baseline were reported. A Partial Mayo Score (mayo score without endoscopy) graded from 0 (normal or inactive disease) to 9 (severe disease) and calculated as the sum of 3 subscores (stool frequency, rectal bleeding and PGA) with each grading from 0 to 3 with higher scores indicating more severe disease.
Time Frame: Baseline, Weeks 2, 4, 8
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 476 | 122
units on a scale
  Change at Week 2: (n= 464, 121) | -2.1 (0.1) | -1.2 (0.2)
  Change at week 4: (n= 460, 117) | -2.8 (0.1) | -1.6 (0.2)
  Change at week 8: (n= 448, 118) | -3.1 (0.1) | -1.6 (0.2)
Statistical Analysis 1: Comparison: Tofacitinib 10 mg BID vs Placebo BID; At Week 2: The change from baseline was analyzed using mixed effect model with treatment group, prior treatment with antiTNF, steroid use at baseline, geographic region, visit and visit by treatment group all as fixed effects, and participants as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed-Effects Model; Least Square Mean Difference = -0.9, 95% CI 2-sided [-1.3 to -0.5], Standard Error of Mean 0.2
Statistical Analysis 2: Comparison: Tofacitinib 10 mg BID vs Placebo BID; At Week 4: The change from baseline was analyzed using mixed effect model with treatment group, prior treatment with antiTNF, steroid use at baseline, geographic region, visit and visit by treatment group all as fixed effects, and participants as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed-Effects Model; Least Square Mean Difference = -1.1, 95% CI 2-sided [-1.5 to -0.7], Standard Error of Mean 0.2
Statistical Analysis 3: Comparison: Tofacitinib 10 mg BID vs Placebo BID; At Week 8: The change from baseline was analyzed using mixed effect model with treatment group, prior treatment with antiTNF, steroid use at baseline, geographic region, visit and visit by treatment group all as fixed effects, and participants as a random effect; Test type: Superiority or Other; p < 0.0001, Mixed-Effects Model; Least Square Mean Difference = -1.5, 95% CI 2-sided [-1.9 to -1.1], Standard Error of Mean 0.2

10. Secondary Outcome: Change From Baseline in Total Mayo Scores at Week 8
Description: Change in total Mayo scores at Week 8 relative to Baseline was reported. Mayo score is an instrument designed to measure disease activity of UC. It consisted of 4 subscores: stool frequency, rectal bleeding, findings of centrally read flexible proctosigmoidoscopy and PGA, each graded from 0 to 3 with higher scores indicating more severe disease. These scores were summed up to give a total score range of 0 to 12; where higher scores indicating more severe disease.
Time Frame: Baseline, Week 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 10 mg BID | Placebo BID
Number analyzed (Participants) | 476 | 122
units on a scale
  Baseline (n= 472, 121) | 9.0 (1.4) | 9.1 (1.4)
  Change at Week 8 (n= 443, 117) | -3.8 (2.8) | -1.9 (2.5)
Statistical Analysis 1: Comparison: Tofacitinib 10 mg BID vs Placebo BID; The change from Baseline at Week 8 was analyzed using an analysis of covariance (ANCOVA) model with treatment group, prior treatment with anti-TNF, steroid use at baseline and geographic region as factors and baseline as a covariate based on the observed-case data; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Square Mean Difference = -1.9, 95% CI 2-sided [-2.5 to -1.4], Standard Error of Mean 0.3

ADVERSE EVENTS:
Time Frame: Baseline up to Day 98
Description: The same event may appear as both an adverse event (AE) and an serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Tofacitinib 10 mg BID | Tofacitinib 15 mg BID | Placebo BID
Serious Adverse Events (participants affected / at risk) | 16/476 | 0/16 | 5/122
Other Adverse Events (participants affected / at risk) | 148/476 | 12/16 | 38/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib 10 mg BID (N=476) | Tofacitinib 15 mg BID (N=16) | Placebo BID (N=122)
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 5 | 0 | 2
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0
Febrile infection (Infections and infestations) | 1 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Vulva cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Aortic dissection (Vascular disorders) | 1 | 0 | 0
Temporal arteritis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib 10 mg BID (N=476) | Tofacitinib 15 mg BID (N=16) | Placebo BID (N=122)
Anaemia (Blood and lymphatic system disorders) | 11 | 1 | 6
Colitis ulcerative (Gastrointestinal disorders) | 6 | 1 | 3
Flatulence (Gastrointestinal disorders) | 2 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 15 | 1 | 5
Fatigue (General disorders) | 10 | 1 | 4
Pyrexia (General disorders) | 14 | 1 | 3
Folliculitis (Infections and infestations) | 9 | 1 | 0
Gastroenteritis (Infections and infestations) | 7 | 1 | 2
Nasopharyngitis (Infections and infestations) | 34 | 3 | 9
Sinusitis (Infections and infestations) | 2 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 15 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 12 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
Headache (Nervous system disorders) | 37 | 0 | 8
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 1 | 1 | 1
Dysuria (Renal and urinary disorders) | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 10 | 3 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 1 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.